CLINICAL TRIAL: NCT05037591
Title: Effect of Sea Grapes-antioxidants Extract in Obese Men
Brief Title: Effect of Sea Grapes-antioxidants Extract in Obese Men : 4 Weeks Randomized-Double Blind Controlled Trial
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: State Islamic University of Sunan Kalijaga Yogyakarta (Other)
Responsible Party: Principal Investigator, Fahrul Nurkolis, Principal Investigator, State Islamic University of Sunan Kalijaga Yogyakarta
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7171011P321452021061500018
Record Dates: First submitted 2021-08-24; First posted 2021-09-08 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Obesity; Aging; Diabetes
Keywords: Obesity; Aging; Functional Food; Diabetes; Dyslipidemia
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Dyslipidemias

STUDY DESIGN:
Intervention Model Description: The study was a 4-week, randomized, double-blind, placebo-controlled clinical trial. Evaluation during the initial visit includes physical examination in the form of Body Mass Index based on Asia-Pacific guidelines and blood parameter screening tests in the form of blood glucose, triglycerides, high-density lipoprotein (HDL), low-density lipoprotein (LDL) and total cholesterol, and PGC-1α were performed on all participants within 1 week of the initial screening. A random number between 1 and 70 was generated for each subject and registered participants were scheduled for their first visit and randomly assigned to the sea grape extract group (n=35) or placebo (n=35). Sea grape extract/placebo tablets/capsules were given to participants every 1 week (1 day of consumption per oral) 15 Minutes before eating (According to the diabetes drug guidline consumtion).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (40):
- placebo A (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo B (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo C (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo D (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo E (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo F (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo G (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo H (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo I (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo J (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo K (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo L (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo M (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo N (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo O (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo P (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo Q (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo R (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo S (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- placebo T (Placebo Comparator): placebo lactose powder (1.68 g/70kg BW day-1) or placebo tablets were given to this group/arms
  Interventions: Drug: Placebo
- sea grape extract A (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract B (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract C (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract D (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract E (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract F (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract G (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract H (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract I (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract J (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract K (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract L (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract M (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract N (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract O (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract P (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract Q (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract R (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract S (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW
- sea grape extract T (Experimental): given sea grape extract 1.68 g/70kg BB day-1 were given to this group/arms
  Interventions: Drug: Sea grapes extract 1.68 g/70kg BW

INTERVENTIONS:
Drug: Sea grapes extract 1.68 g/70kg BW — Contains antioxidants 45.66 ± 0.55% and Caulerpin. Sea grapes are usually consumed raw without any indication of poisoning.
  Arms: sea grape extract A; sea grape extract B; sea grape extract C; sea grape extract D; sea grape extract E; sea grape extract F; sea grape extract G; sea grape extract H; sea grape extract I; sea grape extract J; sea grape extract K; sea grape extract L; sea grape extract M; sea grape extract N; sea grape extract O; sea grape extract P; sea grape extract Q; sea grape extract R; sea grape extract S; sea grape extract T
Drug: Placebo — placebo lactose powder (1.68 g/70kg BW day-1).
  Arms: placebo A; placebo B; placebo C; placebo D; placebo E; placebo F; placebo G; placebo H; placebo I; placebo J; placebo K; placebo L; placebo M; placebo N; placebo O; placebo P; placebo Q; placebo R; placebo S; placebo T

SUMMARY:
Doses of 150 mg/kg BW (30 mg/200g BW) sea grape extract in a previous pre-clinical trial, showed that it could improve blood glucose, total cholesterol and serum PGC-1 levels in rats fed a diet high in fat and cholesterol. In addition, you also have hepatoprotective activity (aka non-toxic) in diabetic mice. Previous research, is an in vivo (Pre-clinical) study that has not represented the benefits or efficacy of sea grape extract on variables tested in humans. Therefore, this clinical trial was conducted to support the effect of sea grape extract-antioxidant on blood glucose, total cholesterol, and PGC-1 levels in obese men for 4 weeks using a Randomized-Double Blind Controlled Trial.

DETAILED DESCRIPTION:
The study was a 4-week, randomized, double-blind, placebo-controlled clinical trial followed by a 1-week screening period. Participants who respond to the invitation and meet the entry criteria during the telephone screening interview are scheduled for the initial visit. Evaluation during the initial visit includes physical examination in the form of BMI (Body Mass Index) based on Asia-Pacific guidelines and blood parameter screening tests in the form of blood glucose, triglycerides, high-density lipoprotein (HDL), low-density lipoprotein (LDL) and total cholesterol, and PGC-1α were performed on all participants within 1 week of the initial screening. A random number between 1 and 70 was generated for each subject and registered participants were scheduled for their first visit and randomly assigned to the sea grape extract group (n=35) or placebo (n=35). Sea grape extract/placebo tablets/capsules were given to participants every 1 week (1 day of consumption per oral) 15 Minutes before eating (According to the diabetes drug guidline consumtion).

During the 4-week intervention period, participants were asked to continue their usual diet and not to consume functional foods or other dietary supplements. Anthropometry (BMI), Waist Hip Ratio (WHR) , blood parameters, urine profile (Marker of toxicity), and nutrient intake of both groups were measured before and after the intervention period. During the trial phase, all participants were instructed to maintain their normal diet and physical activity. Each week participants were asked to report assessments of side effects or changes in training, lifestyle, or diet; and to evaluate tablet compliance.

Subjects/Participants The study participants were recruited during 2021 at Manado, Republic of Indonesia. A total of 150 participants agreed to participate in the study. Only individuals men who are obese (BMI ≥ 25 kg m-2 and Waist Hip Ratio (WHR) ≥ 0.90) according to Asia-Pacific guidelines and have not been diagnosed with other diseases were included in the study. To meet guidelines for evaluating the efficacy of functional food referring to the Korea Food and Drug Administration (because Indonesia does not yet exist and Koreas belong to one Asian region so used), very obese participants (BMI ≥ 30 kg m-2) were not included in the study.

In total, 70 participants met the research criteria (age 29.98 ± 3.26 year; weight, ..... ± .... kg; BMI, .... ±.... kg m-2) and were randomly divided into two groups (n = 35 each) given sea grape extract 1.68 g/70kg BB day-1) or placebo (1.68 g/70kg BB day-1). The exclusion criteria for this study are as follows: (a) significant weight variation (over 10%) in the last 3 months; (b) a history of cardiovascular disease including arrhythmia, heart failure, or myocardial infarction, diabetes mellitus (DM) and the use of pacemakers; (c) a history of conditions that may interfere with test products or inhibit their absorption such as gastrointestinal diseases (Crohn's disease) or surgeries that have been experienced (caesarean section or enterocele); (d) participation in other clinical trials in the last 2 months; (e) abnormal liver function; (f) a history of kidney disease (eg, acute or chronic renal failure and nephrtic syndrome); (g) undergo antipsychotic drug therapy within the last 2 months; (h) laboratory test results as well as medical or psychological conditions that may interfere with successful participation in research assessed by researchers; (i) a history of alcohol or substance abuse; and (j) allergy or hypersensitivity to any of the ingredients in the test product; (k) is neither a passive nor an active smoker. All participants give written consent before the investigation begins. The research protocol was submitted to the Health Research Ethics Commission (KEPK) of The General Hospital of Education Prof. Dr. RD. Kandou (Manado, Republic of Indonesia) online at http://sim-epk.keppkn.kemkes.go.id. All protocols referred to The Declaration of Helsinki and The Council for International Organizations of Medical Sciences (CIOMS).

Measurement of Efficacy Results A total of 70 participants who met the research criteria were asked to visit the clinic once every 1 week (0th, 1st, 2nd, 3rd, and 4th/last week of the study period) with a total of 5 clinical visits including initial examination. During each visit, the use of the supplement is currently reviewed and symptoms or side effects are noted. During screening visits, demographic and lifestyle information is collected (age, alcohol consumption, and smoking habits). Medical history is taken and urine turbidity tests are carried out.

The following parameters are assessed; Weight, Height, WHR and BMI during each visit. Blood samples were collected after a minimum of 12 hours of fasting during initial screening as well as in the 0, 2nd and 4th weeks of the intervention period to obtain blood glucose profiles, total cholesterol, triglycerides, high-density lipoprotein (HDL), low-density lipoprotein (LDL) and PGC-1α. Blood samples were taken from the arm vein. The arm vein to be punctured is cleaned with 70% alcohol and allowed to dry. A tourniquet is placed on the upper arm to expose and slightly accentuate the veins. The skin is stretched over the vein with the fingers of the left hand so that the vein cannot move. The skin is pierced with a needle and syringe with the right hand until the tip of the needle enters the lumen of the vein. The tourniquet is removed and slowly withdraw the syringe suction until the desired amount of blood is obtained. A 70% alcohol swab is placed over the needle and the syringe and needle are removed. The needle is removed from the syringe and the blood sample is transferred into a vacutainer tube.

Evaluation of Safety and Diet

The safety of the extract is assessed by the following procedure. Urine Test Strips 10 Verify Parameters, Parameters examined are:

* Glucose (50 -100 mg / dl)
* Protein (7.5 - 15 mg / dl)
* pH (5-9)
* Leukocytes (9-15 leu / ul)
* Nitrite (0.05-0.1 mg/ dl)
* Urobilinogen (0.2-1.0 mg / dl)
* Blood (5-10 Ery/ul)
* Ketones (2.5-5 mg/dl)
* Bilirubin (0.4-1.0 mg/ dl)
* Specific Gravity (SG) (1,000-1,030) Test the urine parameters above using Urinalysis 10U Reagent Strips Verify (REF U031-102 exp. 2022-03-05). Pulse rate and blood pressure are measured on each visit after a 5-minute break using intelliVue MP70 (Philips, Netherlands). Personal reports are also recorded at these times. We kept the subjects maintaining their usual diet and activity, and all participants completed diet records on each visit to the clinic during the intervention period to evaluate their energy intake and diet quality. Food intake data were analyzed by a nutritionist (Melvin Junior Tanner, S.Gz).

Statistical Analysis Statistical analysis is performed using SPSS software, version 26 (IBM Corporation). Fixed effects include treatment groups, treatment visits, and interactions between treatment and visit groups. The value p<0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Only individuals men who are obese (BMI ≥ 25 kg m-2) according to Asia-Pacific guidelines
* Waist Hip Ratio (WHR) ≥ 0.90 according to Asia-Pacific guidelines and
* not been diagnosed with other diseases were included in the study.

Exclusion Criteria:

* (a) significant weight variation (over 10%) in the last 3 months;
* (b) a history of cardiovascular disease including arrhythmia, heart failure, or myocardial infarction, diabetes mellitus (DM) and the use of pacemakers;
* (c) a history of conditions that may interfere with test products or inhibit their absorption such as gastrointestinal diseases (Crohn's disease) or surgeries that have been experienced (caesarean section or enterocele);
* (d) participation in other clinical trials in the last 2 months;
* (e) abnormal liver function;
* (f) a history of kidney disease (eg, acute or chronic renal failure and nephrtic syndrome);
* (g) undergo antipsychotic drug therapy within the last 2 months;
* (h) laboratory test results as well as medical or psychological conditions that may interfere with successful participation in research assessed by researchers;
* (i) a history of alcohol or substance abuse; and
* (j) allergy or hypersensitivity to any of the ingredients in the test product;
* (k) is neither a passive nor an active smoker.
* All participants give written consent before the investigation begins.

Ages: 19 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Peroxisome proliferator-activated receptor (PPAR)-γ coactivator 1 alpha (PGC-1α) Levels "change" is being assessed | Change from Baseline PGC-1α Levels at 4th weeks of the intervention period
  Evaluate PGC-1α level in pg/dL
Total Cholesterol "change" is being assessed | Change from Baseline Total Cholesterol at 4th weeks of the intervention period
  Evaluate total Cholesterol level in mg/dL
Blood Glucose "change" is being assessed | Change from Baseline Blood Glucose at 4th weeks of the intervention period
  Evaluate total blood sugar level in mg/dL

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Change from Baseline Body Mass Index (BMI) at 4th weeks of the intervention period
  Body Mass Index (BMI) weight and height will be combined to report BMI in kg/m^2
Triglycerides | Change from Baseline Triglycerides Levels at 4th weeks of the intervention period
  Triglycerides in mg/dL
high-density lipoprotein (HDL) | Change from Baseline high-density lipoprotein (HDL) Levels at 4th weeks of the intervention period
  high-density lipoprotein (HDL) in mg/dL
low-density lipoprotein (LDL) | Change from Baseline low-density lipoprotein (LDL) Levels at 4th weeks of the intervention period
  low-density lipoprotein (LDL) in mg/dL
Body Weight | Change from Baseline Body Weight at 4th weeks of the intervention period
  Weight in kilograms (kg)
Body Height | Change from Baseline Body Height at 4th weeks of the intervention period
  Height in meters (M)
waist-to-hip ratio (WHR) | Change from Baseline waist-to-hip ratio (WHR) at 4th weeks of the intervention period
  This is calculated as waist measurement divided by hip measurement (W⁄H). For example, a person with a 30" (76 cm) waist and 38" (97 cm) hips has a waist-hip ratio of about 0.78.

CONTACTS AND LOCATIONS:
Overall Officials: Fahrul Nurkolis, Principal Investigator — UIN Sunan Kalijaga Yogyakarta
Locations (1):
- Fahrul Nurkolis, Manado, North Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Only measurement data with anonymized names will be shared.
Supporting Information: SAP, CSR
Time Frame: After research
Access Criteria: repository

REFERENCES:
- See also: Related Info — https://www.elsevier.com/books/evaluation-of-drug-activities/laurence/978-1-4832-2845-7
- See also: Related Info — https://doi.org/10.12688/f1000research.54952.1

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/91/NCT05037591/Prot_SAP_ICF_000.pdf